CLINICAL TRIAL: NCT06859307
Title: Intra-Abdominal Instillation Of Fresh Frozen Plasma Versus Corticosteroids In Prevention Of Recurrent Attacks Of Adhesive Intestinal Obstruction: A 2 Years' Experience Clinical Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Reham Zakaria Mohamed Ahmed, lecturer of general surgery, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #1109\25-Feb-2025
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-02

CONDITIONS: Adhesive Peritoneal Band
Keywords: adhesions; corticosteroids; fresh frozen plasma
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group I: adhesive intestinal obstruction (Active Comparator)
  Interventions: Procedure: intra-abdominal instillation of corticosteroids
- group II: adhesive intestinal obstruction (Active Comparator)
  Interventions: Procedure: intra-abdominal instillation of fresh frozen plasma

INTERVENTIONS:
Procedure: intra-abdominal instillation of corticosteroids — after adhesiolysis, peritoneal lavage with diluted corticosteroids will be instillated intra-abdominally
  Arms: group I: adhesive intestinal obstruction
Procedure: intra-abdominal instillation of fresh frozen plasma — after adhesiolysis, peritoneal lavage with diluted FFP will be instillated intra-abdominally
  Arms: group II: adhesive intestinal obstruction

SUMMARY:
Adhesive Intestinal obstruction is an inevitable complication of abdominal surgery with significant morbidity associated with poor quality of life and predispose to repeated hospitalization. Most of them (73% - 90%) can be managed conservatively.Despite advances in surgery, 15to 30% require surgical intervention primarily or due to failure of conservative management. Because of the nature of the disease recurrence has been estimated to be 30%.Many attempts to prevent formation of postoperative adhesions have been tried. In this trial, we will study the effect of corticosteroids and FFP in prevention of adhesive small bowel obstruction recurrence for follow up of 2 years duration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with attacks of adhesive intestinal obstruction

Exclusion Criteria:

* Associated abdominal malignancy, patients with adhesive IO who respond to conservative treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
intestinal obstruction | from 1 day to 2 years post operative
  intestinal obstruction is detected if the patient had constipation and vomiting with ultrasound showing dilated bowel and to and fro movement and the plain erect shows multiple air fluid levels
bowel injury | from 1 day to 2 years post operative
  bowel injury will be detected if intestinal contents present in the drain or wound
wound infection | from 1 day to 2 weeks post-operative
  wound infection is detected if there is pus in the drain or wound

SECONDARY OUTCOMES:
age | from 2 to 3 days before surgery
  age will be recorded in years
sex | from 2 to 3 days before surgery
  The sex of the patient will be recorded (male or female)

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of Medicine, Zagazig, Sharqia Province
  - Zagazig University Hospitals, Zagazig, zagazig

IPD SHARING:
Plan to Share IPD: Undecided
data will be available on demand by contacting the principle investigator